CLINICAL TRIAL: NCT05591417
Title: Comparison of Dexmedetomidine and Dexamethasone as Adjuvant to Bupivacaine in Ultrasound-guided Bilevel Erector Spinae Plane Block in Modified Radical Mastectomy
Brief Title: Dexmedetomidine vs Dexamethasone as Adjuvant to Bupivacaine in Bilevel Erector Spinae Plane Block in Breast Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Assistant professor of Anesthesia and Pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP2207-30110
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Dexamethasone; Dexmedetomidine; Morphine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intravenous morphine (Active Comparator): Patients will receive intravenous morphine 0.1 mg/kg
  Interventions: Drug: Intravenous morphine
- Bilevel erector spinae plane block (Experimental): Patients will receive erector spinae plane block at 2 levels
  Interventions: Procedure: Bilevel Erector spinae plane block
- Bilevel erector spinae plane block with dexamethasone (Experimental): Patients will receive erector spinae plane block at 2 levels with dexamethasone
  Interventions: Procedure: Bilateral Erector spinae plane block with dexamethasone
- Bilevel erector spinae plane block with dexmedetomidine (Experimental): Patients will receive erector spinae plane block at 2 levels with dexmedetomidine
  Interventions: Procedure: Bilateral Erector spinae plane block with dexmedetomidine

INTERVENTIONS:
Procedure: Bilevel Erector spinae plane block — Patients will receive bilevel erector spinae plane block with bupivacaine
  Other Names: BileveL ESPB
  Arms: Bilevel erector spinae plane block
Procedure: Bilateral Erector spinae plane block with dexamethasone — Patients will receive bilevel erector spinae plane block with bupivacaine and dexamethasone
  Other Names: Bilevel ESPB with dexamethasone
  Arms: Bilevel erector spinae plane block with dexamethasone
Procedure: Bilateral Erector spinae plane block with dexmedetomidine — Patients will receive bilevel erector spinae plane block with bupivacaine and dexmedetomidine
  Other Names: Bilevel ESPB with dexmedetomidine
  Arms: Bilevel erector spinae plane block with dexmedetomidine
Drug: Intravenous morphine — Intravenous morphine 0.1 mg/kg
  Other Names: Morphine
  Arms: Intravenous morphine

SUMMARY:
High percent of patients experience chronic pain following breast cancer surgeries thus proper perioperative pain control is crucial to lessen the incidence of such pain. Several techniques are adopted to control perioperative pain, these techniques include drugs as opioids and adjuvants as well as regional blocks. Erector spinae plane block is a regional technique that is used efficiently to control perioperative pain during and following breast cancer surgeries.

DETAILED DESCRIPTION:
High percent of patients experience chronic pain following breast cancer surgeries thus proper perioperative pain control is crucial to lessen the incidence of such pain. Several techniques are adopted to control perioperative pain, these techniques include drugs as opioids and adjuvants as well as regional blocks. Erector spinae plane block is a regional technique that is used efficiently to control perioperative pain during and following breast cancer surgeries. Adding adjuvant drugs as dexmedetomidine or dexamethasone can augment the local anesthetic effect for the regional block used.

ELIGIBILITY:
Inclusion Criteria:

* Female patients scheduled for Modified Radical Mastectomy MRM
* Physical status ASA II, III.
* Age (18-65) years
* Body mass index (BMI): (20-35) kg/m2.

Exclusion Criteria:

* Patient refusal.
* Age <18 years or >65 years.
* BMI <20 kg/m2 and >35 kg/m2.
* Known sensitivity or contraindication to drug used in the study (local anaesthetics, opioids, dexamethasone, dexmedetomedine).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 68 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption in the first 24 hours postoperatively. | First 24 hours postoperatively
  Assessment of total postoperative morphine consumption

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Assistant Professor of Anesthesia and Pain Management, National Cancer Institute, Cairo University
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt